CLINICAL TRIAL: NCT00730353
Title: A Phase II Study of Sunitinib Malate (Sutent®) With Paclitaxel (Taxol®) in Patients With Advanced Esophageal Cancer
Brief Title: Sutent + Taxol for Advanced Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Nasser Hanna, M.D., Professor, IU School of Medicine, Hoosier Cancer Research Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GI06-112
Record Dates: First submitted 2008-08-04; First posted 2008-08-08 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Sunitinib; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Treatment will be administered on an outpatient basis. Chemotherapy will be administered in a 28-day treatment cycle. The 28 days of treatment with paclitaxel and sunitinib malate (plus the time required to recover if toxicity is encountered) is defined as a cycle.
  * Paclitaxel 90 mg/m2 IV on days 1, 8 and 15.
  * Sunitinib malate 37.5 mg orally, daily. After 4 cycles, paclitaxel will be discontinued and patients will continue on sunitinib malate until disease progression, unacceptable toxicity, or physician discretion.
  Interventions: Drug: Sunitinib malate; Drug: Paclitaxel

INTERVENTIONS:
Drug: Sunitinib malate — Sunitinib malate 37.5 mg orally, daily
Drug: Paclitaxel — Paclitaxel 90 mg/m2 IV on days 1, 8 and 15.

SUMMARY:
Paclitaxel is known to be active as a single and combination agent in esophageal cancer, and has also been demonstrated to have anti-angiogenic properties in weekly dosing regimens. Sunitinib malate is an anti-angiogenic drug with the potential to improve responses when combined with chemotherapy, as demonstrated with other regimens in similar settings. We believe that the combination of paclitaxel and sunitinib malate offer great promise in the treatment of advanced esophageal cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

Treatment will be administered on an outpatient basis. Chemotherapy will be administered in a 28-day treatment cycle. The 28 days of treatment with paclitaxel and sunitinib malate (plus the time required to recover if toxicity is encountered) is defined as a cycle.

* Paclitaxel 90 mg/m2 IV on days 1, 8 and 15.
* Sunitinib malate 37.5 mg orally, daily.

After 4 cycles, paclitaxel will be discontinued and patients will continue on sunitinib malate until disease progression, unacceptable toxicity, or physician discretion.

Performance Status: ECOG (Eastern Cooperative Oncology Group) performance status 0 to 2

Life expectancy: Not specified

Hematopoietic:

* International Normalized Ratio (INR) < 1.2
* Partial Thromboplastin Time (PTT) < 1.5 x Upper Limit of Normal (ULN)
* Platelets > 100 K/mm3
* Hemoglobin > 8 g/dL
* Absolute Neutrophil Count (ANC) > 1.0 K/mm3

Hepatic:

* Aspartate transaminase (AST) ≤ 2.5 x ULN, or ≤ 5.0 x ULN if the transaminase elevation is due to known liver metastases.
* Alanine transaminase (ALT) ≤ 2.5 x ULN, or ≤ 5.0 x ULN if the transaminase elevation is due to known liver metastases.
* Total bilirubin < 2.0 x ULN

Renal:

* Serum creatinine ≤ 2 x ULN or a calculated creatinine clearance (using Cockcroft-Gault formula) > 50 cc/min

Cardiovascular:

* No history of unstable angina, myocardial infarction, coronary artery bypass grafting surgery within 12 months prior to registration for protocol therapy. Patients may be on anti-anginal medications, but must be stable on those medications for at least 6 months.
* No history of New York Heart Association class II or greater congestive heart failure.

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrent or metastatic esophageal or gastro-esophageal junction squamous cell or adenocarcinoma
* Measurable or evaluable disease per RECIST within 28 days prior to being registered on protocol therapy.
* No more than one prior chemotherapy regimen for locally advanced or metastatic disease is allowed.
* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age > 18 years.
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) while on treatment and for 3 month period thereafter.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy. Subjects are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* Females must not be breastfeeding.
* Must be willing to comply with study and follow up procedures.

Exclusion Criteria:

* No history of inadequately controlled hypertension (Systolic Blood Pressure > 150 or Diastolic Blood Pressure > 100) on a standard regimen of antihypertensive therapy.
* No prior treatment with vascular endothelial growth factor (VEGF) inhibitor, epidermal growth factor receptor (EGFR) inhibitor, or other anti-angiogenic agent.

No serious, non-healing wound, ulcer, or bone fracture.

* No history of or current hemoptysis.
* No history of transient ischemic attack (TIA) or stroke within 12 months prior to registration for protocol therapy.
* No evidence of bleeding diathesis, coagulopathy, prolonged INR or PTT.
* No chronic anti-coagulation treatment.
* No history of central nervous system or brain metastases.
* No history of any major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to registration for protocol therapy, or anticipation of need for major surgical procedure during the course of protocol therapy.
* No history of any minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to registration for protocol therapy.
* No history of clinically significant peripheral neuropathy, i.e., Grade > 3 neuromotor or neurosensory toxicity as defined by NCI CTCAE v 3.0.
* No known history of adrenal insufficiency documented by adrenocorticotropic hormone (ACTH) stimulation testing.
* No prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 450 msec), obtained within 28 days prior to being registered for protocol therapy.
* No other active cancers
* No clinically significant infections as judged by the treating investigator.
* No history of a seizure disorder.
* No known history of hypersensitivity to paclitaxel.
* No CYP3A4 inducers and inhibitors allowed within 14 days prior to registration on protocol therapy and while receiving the protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Cancer Research Network
Locations (15):
- United States (15):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - IN Onc/Hem Associates, Indianapolis, Indiana
  - Indiana University Simon Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Horizon Oncology Center, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Monroe Medical Associates, Munster, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Providence Medical Group, Terre Haute, Indiana
  - Ireland Cancer Center - University Hospitals of Cleveland, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmitt JM, Sommers SR, Fisher W, Ansari R, Robin E, Koneru K, McClean J, Liu Z, Tong Y, Hanna N. Sunitinib plus paclitaxel in patients with advanced esophageal cancer: a phase II study from the Hoosier Oncology Group. J Thorac Oncol. 2012 Apr;7(4):760-3. doi: 10.1097/JTO.0b013e31824abc7c. PMID 22425927
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial opened to accrual November 2008; opened at both community and academic performance sites.
Pre-assignment Details: This trial was limited to patients with advanced esophageal cancer.
Groups:
- Paclitaxel and Sutinib Malate: Treatment will be administered on an outpatient basis. Chemotherapy will be administered in a 28-day treatment cycle. The 28 days of treatment with paclitaxel and sunitinib malate (plus the time required to recover if toxicity is encountered) is defined as a cycle.
  * Paclitaxel 90 mg/m2 IV on days 1, 8 and 15.
  * Sunitinib malate 37.5 mg orally, daily. After 4 cycles, paclitaxel will be discontinued and patients will continue on sunitinib malate until disease progression, unacceptable toxicity, or physician discretion.
Period: Overall Study
Arm/Group | Paclitaxel and Sutinib Malate
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel and Sutinib Malate
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 59.5 [40 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 28
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  Participants
    ECOG PS 0 | 15
    ECOG PS 1 | 11
    ECOG PS 2 | 2
Tumor Site [Number; unit: participants]
  Esophagus | 22
  Gastroesophageal Junction | 6
Histology [Number; unit: participants]
  Adenocarcinoma | 26
  Squamous cell carcinoma | 2
Prior Treatment [Number; unit: participants]
  Yes | 11
  No | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate at 24 Weeks
Description: To determine the rate of non-progressive disease at 24 weeks from the first dose of the combination of sunitinib malate and paclitaxel in advanced esophageal carcinoma, where progression is defined as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 24 weeks
Population: Intent to treat - all enrolled participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel and Sutinib Malate
Number analyzed (Participants) | 28
percentage of participants | 25 [12 to 42]

2. Secondary Outcome: Response Rate
Description: To determine the response rate for the combination of sunitinib malate and paclitaxel in advanced esophageal carcinoma per RECIST criteria.
Time Frame: 6 months
Population: Evaluable patients, as previously defined.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel and Sutinib Malate
Number analyzed (Participants) | 23
percentage of participants | 13 [3 to 25]

3. Secondary Outcome: Overall Survival
Description: To determine the one year overall survival rate for the combination of sunitinib malate and paclitaxel in advanced esophageal carcinoma
Time Frame: 12 months
Population: All participants on an intent-to-treat basis
Measure: Median (90% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel and Sutinib Malate
Number analyzed (Participants) | 28
percentage of participants | 20 [9 to 34]

4. Secondary Outcome: Progression-Free Survival
Description: To determine the time to progression for the combination of sunitinib malate and paclitaxel in advanced esophageal carcinoma per RECIST criteria.
Time Frame: 12 months
Population: Intention-to-treat patients
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Paclitaxel and Sutinib Malate
Number analyzed (Participants) | 28
Days | 112 [54 to 150]

5. Secondary Outcome: Toxicity Profile
Description: Determine the most frequent toxicities associated with the treatment regimen, per the CTCAE version 3 (Common Toxicity Criteria for Adverse Events) criteria.
Time Frame: 16 months
Measure: Number; unit: instances of adverse event
Arm/Group | Paclitaxel and Sutinib Malate
Number analyzed (Participants) | 28
instances of adverse event
  Leukopenia/neutropenia: Grade 3/4 | 7
  Anemia: Grade 3/4 | 5
  Thrombocytopenia | 1
  Febrile Neutropenia | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Paclitaxel and Sutinib Malate
Serious Adverse Events (participants affected / at risk) | 14/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Sutinib Malate (N=28)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (4)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (2)
DEATH NOT ASSOCIATED WITH CTCAE TERM / DEATH NOS (General disorders) | 1 (1)
DERMATOLOGY/SKIN - OTHER (Skin and subcutaneous tissue disorders) | 1 (1)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FISTULA, GI / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
HEMOGLOBIN (Blood and lymphatic system disorders) | 1 (1)
HEMORRHAGE, GI / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, GI / STOMACH (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, GI / UPPER GI NOS (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE/BLEEDING - OTHER (General disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BONE (OSTEOMYELITIS) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FLUTTER (Cardiac disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Sutinib Malate (N=28)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 3 (3)
ALKALINE PHOSPHATASE (Investigations) | 9 (16)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 2 (2)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 4 (6)
AMYLASE (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 20 (24)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 2 (2)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 8 (15)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 2 (3)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 12 (19)
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 (19)
CYSTITIS (Renal and urinary disorders) | 1 (1)
CYTOKINE RELEASE SYNDROME/ACUTE INFUSION REACTION (Immune system disorders) | 2 (4)
DEHYDRATION (Gastrointestinal disorders) | 3 (4)
DIARRHEA (Gastrointestinal disorders) | 12 (27)
DIZZINESS (Nervous system disorders) | 4 (4)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 3 (3)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSPHAGIA (DIFFICULTY SWALLOWING) (Gastrointestinal disorders) | 13 (18)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 13 (18)
EDEMA: LIMB (Blood and lymphatic system disorders) | 3 (3)
EDEMA: TRUNK/GENITAL (Blood and lymphatic system disorders) | 1 (1)
ENDOCRINE - OTHER (Endocrine disorders) | 1 (1)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 23 (52)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
FEVER (General disorders) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 3 (3)
FISTULA, GI / ESOPHAGUS (Gastrointestinal disorders) | 2 (2)
FLUSHING (Skin and subcutaneous tissue disorders) | 2 (2)
GASTROINTESTINAL - OTHER (Gastrointestinal disorders) | 1 (1)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 7 (12)
GLUCOSE, SERUM-LOW (HYPOGLYCEMIA) (Investigations) | 1 (1)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 13 (18)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 12 (18)
HEMOGLOBIN (Blood and lymphatic system disorders) | 19 (40)
HEMORRHAGE, GI / VARICES (RECTAL) (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 4 (5)
HEMORRHAGE/BLEEDING - OTHER (General disorders) | 2 (3)
HEMORRHOIDS (Gastrointestinal disorders) | 1 (1)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
HOT FLASHES/FLUSHES (Endocrine disorders) | 3 (4)
HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 2 (2)
HYPOTENSION (Cardiac disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / MUCOSA (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / PENIS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SINUS (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AIRWAY NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / WOUND (Infections and infestations) | 1 (1)
INJECTION SITE REACTION/EXTRAVASATION CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
INR (INTERNATIONAL NORMALIZED RATIO OF PROTHROMBIN TIME) (Surgical and medical procedures) | 1 (1)
INSOMNIA (General disorders) | 12 (18)
LEFT VENTRICULAR DIASTOLIC DYSFUNCTION (Cardiac disorders) | 1 (1)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 5 (21)
LIPASE (Investigations) | 1 (1)
LYMPHEDEMA-RELATED FIBROSIS (Blood and lymphatic system disorders) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (2)
METABOLIC/LABORATORY - OTHER (Investigations) | 3 (3)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (1)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 8 (10)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 10 (12)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ANUS (Surgical and medical procedures) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 5 (6)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ESOPHAGUS (Gastrointestinal disorders) | 2 (4)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 2 (2)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 5 (6)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 1 (1)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 16 (24)
NEUROLOGY - OTHER (Nervous system disorders) | 2 (2)
NEUROPATHY: MOTOR (Nervous system disorders) | 1 (1)
NEUROPATHY: SENSORY (Nervous system disorders) | 12 (14)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 11 (32)
OBSTRUCTION/STENOSIS OF AIRWAY / BRONCHUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 9 (15)
PAIN / ANUS (Gastrointestinal disorders) | 1 (3)
PAIN / BACK (General disorders) | 10 (12)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 3 (5)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 5 (5)
PAIN / DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 1 (1)
PAIN / ESOPHAGUS (Gastrointestinal disorders) | 2 (2)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 5 (8)
PAIN / HEAD/HEADACHE (General disorders) | 5 (5)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN / ORAL-GUMS (Gastrointestinal disorders) | 1 (1)
PAIN / RECTUM (Gastrointestinal disorders) | 1 (1)
PAIN / STOMACH (Gastrointestinal disorders) | 1 (1)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 2 (3)
PAIN / TUMOR PAIN (General disorders) | 1 (1)
PAIN - OTHER (General disorders) | 4 (5)
PLATELETS (Blood and lymphatic system disorders) | 5 (11)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 2 (4)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 1 (1)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 1 (1)
PTT (PARTIAL THROMBOPLASTIN TIME) (Surgical and medical procedures) | 1 (1)
PULMONARY/UPPER RESPIRATORY - OTHER (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 4 (5)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 2 (2)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 3 (4)
RIGORS/CHILLS (General disorders) | 5 (6)
SALIVARY GLAND CHANGES/SALIVA (Gastrointestinal disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 5 (7)
SWEATING (DIAPHORESIS) (General disorders) | 2 (2)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 5 (8)
THYROID FUNCTION, HIGH (HYPERTHYROIDISM, THYROTOXICOSIS) (Endocrine disorders) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 3 (3)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 8 (12)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 2 (2)
WEIGHT LOSS (General disorders) | 5 (5)

LIMITATIONS AND CAVEATS:
Statistical power is based on 26 evaluable patients; However, all objectives other than the primary objective were based on 23 evaluable patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No